CLINICAL TRIAL: NCT03847324
Title: Physiotherapy and Therapeutic Education on Patients With Pain Catastrophism Scheduled for a Total Knee Arthroplasty: Randomized Clinical Trial
Brief Title: Physiotherapy and Therapeutic Education on Patients With Pain Catastrophism Scheduled for a Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: Hector Beltran-Alacreu, PhD (Unknown)
Responsible Party: Principal Investigator, Marc Terradas Monllor, Marc Terradas-Monllor, Msc, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FISIOPTR-01
Record Dates: First submitted 2019-02-18; First posted 2019-02-20 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Osteo Arthritis Knee; Knee Arthroplasty; Catastrophizing; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Three armed, parallel groups, single blind, unicentric randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (Active Comparator): Group-based preoperative biomedical education, postoperative hospital and home rehabilitation.
  Interventions: Other: Usual Care
- PNE (Experimental): Usual care + Preoperative Pain Neuroscience Education
  Interventions: Other: Pain Neuroscience Education; Other: Usual Care
- Multimodal Physiotherapy (Experimental): Usual care + Preoperative Multimodal physiotherapy
  Interventions: Other: Multimodal Physiotherapy; Other: Usual Care

INTERVENTIONS:
Other: Pain Neuroscience Education — This program is mainly based in "Explain Pain" concept, used in multiple rehabilitation programs. Its aim is to change the subject's pain understanding, teaching them the biological processes underneath the pain construct, as a mechanism to reduce itself and its related maladaptive thoughts and behaviors.
  Other Names: Pain Education
  Arms: PNE
Other: Multimodal Physiotherapy — This intervention will be divided in pain neuroscience education, orthopedic manual therapy and therapeutic exercise.
  Arms: Multimodal Physiotherapy
Other: Usual Care — Usual care will be divided in: preoperative biomedical group-based education, postoperative hospital rehabilitation and home-based postoperative physiotherapy.

SUMMARY:
The purpose of this study is to test whether adding a treatment using pain neuroscience education (PNE) and multimodal physiotherapy to usual care, in subjects with knee osteoarthritis and pain catastrophizing, who are scheduled for a total knee arthroplasty (TKA), is more effective than only usual care. There is a high evidence level of different systematic reviews, which support the efficacy of physiotherapy treatments combined with behavioural/educational techniques aimed to reduce pain catastrophism, pain and disability in other pathologies. The primary aim of that kind of interventions is to help the subjects to reconceptualise its own pain understanding and its role on the recovery process, as well as promoting an increase of activity and encourage the subject to resume its usual activity instead of continuing to avoid it.

DETAILED DESCRIPTION:
The prevalence of TKA has increased dramatically during the last two decades, its popularity can be attributed to its evident success regarding pain improvement, deformity correction and disability reduction in knee osteoarthritis subjects. However, only a third of the patients report no functional problems after surgery, the 20% of then are unsatisfied with its functional skills and around a 20% are experiencing pain, high disability degrees and a significant quality of life reduction. This results cannot be fully explained by mechanical processes, surgical procedures or surgery variations, but it seems to be related to other psychological aspects. Chronic pain subjects often develop maladaptive thoughts and behaviours (i.e. pain catastrophism, Kinesiophobia, activity avoidance) which contribute to make the subject suffer physically as well as emotionally, and affect on the intensity and persistency of pain.

Although many psychosocial factors have been studied, pain catastrophism has emerged as one of the most important predictors for persistent pain after a total knee arthroplasty, as well as its severity and duration, that's why it is getting more importance when it comes to study chronic pain in this subjects. Reducing pain catastrophism has become a key factor to determine the success in the rehabilitation of some maladies accompanied by pain, considering that its reduction has been associated with the clinical improvement of pain itself. It has been observed that treatments using psychological and psychosocial interventions, therapeutic education and coping skills training, or physical therapy and therapeutic exercise, are effective techniques to reduce pain catastrophism. Nevertheless, it's still necessary to determine whether the maladaptive pain related thoughts approach, using physical therapy and behavioural techniques, are able to reduce the risk of suffering postoperative chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* To have sufficient Spanish or Catalan reading, writing and speaking skills to comprehend all explanations and to complete the assessment tools.
* Be able to provide the informed consent.
* Be scheduled to undergo in a total knee arthroplasty.
* Primary knee osteoarthritis diagnosis.
* Score more than 20 points in the Pain Catastrophizing Scale (PCS).
* Score more than 4 over 10 on pain Visual Analogue Scale (VAS)
* Patients older than 18 years old.

Exclusion Criteria:

* Patients scheduled to undergo in a total knee arthroplasty because of prostheses replacement, tumor, infection or fracture.
* Patients scheduled to undergo in a bilateral total knee arthroplasty.
* Patients that will need another total knee or hip replacement surgery in less than a year regarding the current intervention.
* Patients scheduled for unicompartmental knee arthroplasty.
* Patients with other pathologies with characteristic features of a central sensitization. (i.e. Fibromyalgia)
* Co-existing other inflammatory or rheumatic conditions (i.e. rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus or ankylosing spondylitis)
* Co-existing other mental condition and/or major depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Pain. Changes from baseline 6 months post-surgery. | Baseline, 2 weeks before surgery, 1, 3 and 6 months after surgery.
  Participants will be asked to rate their pain intensity on a horizontal 100-mm Visual Analogue Scale (VAS), ranging from 0 = no pain to 100 = worst imaginable pain. The VAS is a valid and reliable instrument compared with other pain rating scales, and has been well established in clinical practice and research for measuring pain levels in arthritis populations.

SECONDARY OUTCOMES:
Range of Motion | Baseline, 2 weeks before surgery, 1, 3 and 6 months after surgery.
  Goniometric assessments of knee will be carried out to assess flexion and extension range of motion.
Walking Speed | Baseline, 2 weeks before surgery, 1, 3 and 6 months after surgery.
  4 Meters Walking Test (4MWT) will be used to evaluate patient's walking speed.
Function | Baseline, 2 weeks before surgery, 1, 3 and 6 months after surgery.
  30-Second Chair Stand Test (30sCST) will be use to evaluate patient's functionality on standing, because it is a well-recognized test to detect early declines in functional independence.
Dynamic Balance | Baseline, 2 weeks before surgery, 1, 3 and 6 months after surgery.
  Y Balance Test (YBT) will be use to evaluate patient's dynamic balance.
Disability / Limitation | Baseline, 2 weeks before surgery, 1, 3 and 6 months after surgery.
  Western Ontario and McMaster University Osteoarthritis Index (WOMAC) (Spanish version) will be used to assess patient´s physical function. This questionnaire can be completed in less than 5 minutes. It's a widely used, reliable, valid and responsive measure of outcome in people with osteoarthritis of the hip or knee.
Health-related Quality of Life | Baseline, 2 weeks before surgery, 1, 3 and 6 months after surgery.
  The spanish version of the Euro Quality of Life 5D-5L (EQ-5D-5L) was used to assess the health related quality of life (HRQL).(10) The EQ-5D-5L consists in two pages: the first one is based on a descriptive system that defines health in terms of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five response categories: no problems, slight problems, moderate problems, severe problems, extreme problems.(10) A health state is composed by taking one level for each dimension, and a preference-based scoring function is used to convert the descriptive system to a summary index score (ranging from states worse than dead <0 to full health 1).
Pain Catastrophism | Baseline, 2 weeks before surgery, 1, 3 and 6 months after surgery.
  The Spanish version of Pain Catastrophizing Scale (PCS) was used to asses thoughts and feelings related to pain experiences.(9) The PCS is a 13 item self-administered questionnaire composed of 3 subscales: rumination, magnification and helplessness. The PCS uses a 5-point Likert scale with responses ranging from 0 = not at all to 4 = all the time. Overall scores range from 0 to 52 points, the higher the score, the higher is the pain catastrophism level.
Depression and anxiety | Baseline, 2 weeks before surgery, 1, 3 and 6 months after surgery.
  Participants will be asked to complete the Hospital Anxiety and Depression Scale (HADS) (Spanish version) will be used. The HADS is a 14 item self-administered questionnaire comprised of 2 subscales: depression and anxiety, both composed with 7 items. Each item use a 4-point Likert scale with responses ranging from 0 to 4. Overall scores range from 0 to 21 points for each subscales, and final score is presented using each subscale scores separately. The higher the score, the higher are the anxiety or depression levels.
Kinesiophobia | Baseline, 2 weeks before surgery, 1, 3 and 6 months after surgery.
  Participants will be asked to complete the Tampa Scale for Kinesiophobia (TSK-11) (Spanish version). TSK-11 is a 11 item self-administered questionnaire used to assess the pain-related fear of movement. The TSK-11 uses a 4-point Likert scale with responses ranging from 1 = totally disagree, to 4 = totally agree. Overall scores range from 11 to 44 indicating a higher degree of pain-related fear of movement when the score is higher.
Self-efficacy | Baseline, 2 weeks before surgery, 1, 3 and 6 months after surgery.
  Participants will be asked to complete the Chronic Pain Self-Efficacy Scale (Spanish version). The Chronic Pain Self-Efficacy Scale is a 19 item self-administered questionnaire used to asses pain-related self-efficacy. It uses a visual analog scale for each item, ranging from 0 = totally uncapable to 10 = totally capable. Overall score ranges from 0 to 190. The higher the score, the higher is the subjects' self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Germans Trias i Pujol, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Terradas-Monllor M, Beltran-Alacreu H, Ochandorena-Acha M, Garcia-Oltra E, Aliaga-Orduna F, Hernandez-Hermoso J. Preoperative Home-Based Multimodal Physiotherapy in Patients Scheduled for a Knee Arthroplasty Who Catastrophize About Their Pain: A Randomized Controlled Trial. J Clin Med. 2025 Jan 5;14(1):268. doi: 10.3390/jcm14010268. PMID 39797350